CLINICAL TRIAL: NCT03955159
Title: Effects of Probiotic Supplementation on Autonomic Nervous System Imbalance and Vascular Changes in Hypertensive Menopausal Women: RANDOMIZED CLINICAL TRIAL
Brief Title: Effects of Probiotic Supplementation in Hypertensive Women on Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Aline Dalmazo, Principal Investigator, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 549019
Record Dates: First submitted 2019-04-15; First posted 2019-05-17 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Systemic Arterial Hypertension; Menopause; Dysbiosis; Autonomic Nervous System Imbalance
MeSH Terms: conditions — Hypertension; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Probiotic supplementation (Experimental): The probiotic is composed of the combination of Lactobacillus acidophilus and Bifidobacterium lactis, at the concentration of 109 CFU. This product presents no known hazards associated with its use. On the contrary, the use of this supplement is associated with a rebalancing of the intestinal microbiota with potential secondary benefits to the reconstitution of the intestinal symbiosis. Patients will receive 1 sachet of 1 gram per day and will be advised to dilute in 100 mL in water at room temperature for administration.
  Interventions: Dietary Supplement: Probiotic supplementation
- Placebo comparator (Placebo Comparator): The placebo that will be used in the present study is maltodextrin, which is a food supplement based on carbohydrate powder.
  Interventions: Dietary Supplement: Probiotic supplementation

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation — The probiotic is composed of the combination of Lactobacillus acidophilus and Bifidobacterium lactis, at the concentration of 109 CFU. This product presents no known hazards associated with its use. On the contrary, the use of this supplement is associated with a rebalancing of the intestinal microbiota with potential secondary benefits to the reconstitution of the intestinal symbiosis. Patients will receive 1 sachet of 1 gram per day and will be advised to dilute in 100 mL in water at room temperature for administration.

SUMMARY:
In postmenopausal women, cardiovascular risk is increased and the mechanisms involving imbalance of the Autonomic Nervous System should be extensively investigated. Recent data suggest a link with intestinal microbiota dysbiosis and probiotic supplementation could be a useful strategy for treating women with increased cardiovascular risk.

DETAILED DESCRIPTION:
After randomization, subjects will be included in their intervention group for a period of three months with initial and final evaluations.

The study will evaluate the effects and possible benefits of probiotic supplementation on the functioning of the Autonomic Nervous System and vascular changes in hypertension in menopausal women.

The intervention groups will be as follows:

1. - Menopausal women with hypertension + Probiotic supplementation
2. - Menopausal women with hypertension + Placebo supplementation

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive
* At least 1 year of menopause
* Sedentary

Exclusion Criteria:

* Smoker
* Use of psychiatric medications
* Cardiovascular events
* Recent surgeries
* Diabetic
* Use of beta blockers

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Autonomic Nervous System | 3 months
  The data will be collected through the system of acquisition of pressure waves in a continuous and non-invasive way by the Finometer® system, through a cuffing installed in the middle finger, taking this signal to an analog-to-digital signal converter. The pulse pressure signal will be acquired at 1000 Hz, continuously and non-invasively, supine (10 minutes) in a quiet environment, with controlled temperature (± 23 ° C) and illumination.
  The collected data will be saved in the software BeatsScope® and LabChart®, from which will be extracted the syistograms for analysis.
  The autonomic nervous system will be assessed at baseline and after 3 months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Claudia Irigoyen, PhD, Study Chair — Instituto de Cardiologia - Fundação Universitária de Cardiologia
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No